CLINICAL TRIAL: NCT07378163
Title: Study on the Preferences for Percutaneous Coronary Intervention Implantation Devices Among Healthcare Providers and Patients With Coronary Artery Disease
Brief Title: Study on the Preferences for PCI Implantation Devices Among Doctors and Patients
Acronym: REC-DEVICEPREF
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the Department of Cardiology, Xijing Hospital
Other Study IDs: REC-DEVICEPREF
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Coronary artery disease; drug-coated balloon; drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Medical staff and patients with CAD
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire regarding the preference of DCB or DES-based PCI among patients with CAD and medical staff

SUMMARY:
The contemporary percutaneous treatment of coronary artery disease typically involves initial lesion preparation with balloon angioplasty, followed by the deployment of a drug-eluting stent (DES) to provide an immediate scaffold and reduce the long-term risk of restenosis. However, stent implantation continues to present notable challenges, primarily due to the metallic scaffold left behind. Compared to DES, drug-coated balloons (DCB) provide a direct release of antiproliferative drugs into the vessel wall, preventing coronary restenosis after angioplasty and limiting the risk of stent-related events. DCBs are an established treatment option for in-stent restenosis and small vessels. However, the REC-CAGEFREE I trial demonstrated that a strategy of DCB angioplasty with rescue stenting did not achieve non-inferiority compared with the intended DES implantation in patients with de novo, non-complex coronary artery disease (CAD), irrespective of vessel diameter.

Previous studies have mainly focused on the efficacy of PCI strategies in reducing adverse event rates, while less attention has been paid to patients' willingness regarding stent implantation. The AHA conducted a systematic review on depression and poor prognosis among patients with acute coronary syndrome (ACS), concluding that health organizations should consider depression as an official risk factor for poor prognosis after ACS. A prior study of patients with coronary artery disease after stent implantation found that their anxiety stemmed primarily from concerns about the stent's long-term effects and its impact on their social interaction. However, data regarding patients' preferences on the selection of DES or DCB is scarce, and whether the psychological impact would differ between DES- or DCB-treated patients is still unknown. This study aimed to investigate the preferences of patients, as well as medical staff, for DES or DCB-based PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute or chronic coronary syndrome who have undergone percutaneous coronary intervention;
2. Patients who can understand the purpose of this trial and are willing to participate in the preference questionnaire.
3. Healthcare providers who treat patients with coronary artery disease.

Exclusion Criteria:

1. Aged < 18 years;
2. Inability to understand the questionnaire or presence of cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare providers and patients with CAD
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum acceptable risk in the trade-off of death | Before discharge
  To avoid permanent metallic stent implantation, the maximum acceptable increase in risk for patients and medical staff in choosing DCB treatment.
Maximum acceptable risk in the trade-off of stroke | Before discharge
  To avoid permanent metallic stent implantation, the maximum acceptable increase in risk for patients and medical staff in choosing DCB treatment.
Maximum acceptable risk in the trade-off of myocardial infarction | Before discharge
  To avoid permanent metallic stent implantation, the maximum acceptable increase in risk for patients and medical staff in choosing DCB treatment.
Maximum acceptable risk in the trade-off of cardiopulmonary resuscitation | Before discharge
  To avoid permanent metallic stent implantation, the maximum acceptable increase in risk for patients and medical staff in choosing DCB treatment.
Maximum acceptable risk in the trade-off of revascularization | Before discharge
  To avoid permanent metallic stent implantation, the maximum acceptable increase in risk for patients and medical staff in choosing DCB treatment.
Maximum acceptable risk in the trade-off of rehospitalization | Before discharge
  To avoid permanent metallic stent implantation, the maximum acceptable increase in risk for patients and medical staff in choosing DCB treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D, Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China